CLINICAL TRIAL: NCT02602171
Title: Virtual Acoustic Localization Experiment for the Evaluation of a Dereverberation Algorithm in Terms of Speech Intelligibility & Localization Performance of Normal Hearing & Hearing Impaired Subjects
Brief Title: Virtual Acoustic Localization Experiment
Acronym: VALEEvE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DN_23_10_15
Record Dates: First submitted 2015-11-04; First posted 2015-11-11 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- dereverberation condition (Experimental): Oldenburger Sentence test, localization test
  Interventions: Other: Oldenburger sentence test, localization test
- reverberation condition (Experimental): Oldenburger Sentence test, localization test
  Interventions: Other: Oldenburger sentence test, localization test

INTERVENTIONS:
Other: Oldenburger sentence test, localization test

SUMMARY:
The present study has the evaluation of a test to measure the localization performance goal . It is about the perception of danger audio signals in everyday listening environments nearby which are reproduced in controlled laboratory conditions. In addition, a dereverberation algorithm regarding speech intelligibility and localization ability is evaluated . The research hypothesis is that the dereverberation of the audio signals can improve speech intelligibility for both normal hearing and hearing-impaired persons. In addition, the binaural dereverberation algorithm should not affect the localization ability in everyday situations.

ELIGIBILITY:
Inclusion Criteria:

* adults , in general healthy (no diagnosis of dementia and/or stroke known), mother tongue: (swiss) german, normal hearing or with hearing aid wearers both sides or with CI support on both sides, symmetrical hearing loss

Exclusion Criteria:

* deviation of inclusion criteria, known fluctuating, rapidly progressive hearing loss, test person is not able to come one time a week to the University Hospital of Zurich or to handle 1-2 hours appointments or is not able to use touchscreen

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Oldenburger sentence test and localization test with 30 subjects | 1 day
  The impact of a dereverberation algorithm for hearing aids and / or cochlear implants will be checked

SECONDARY OUTCOMES:
Differences in localization ability | 1 day
  By VALE (localization test) can differences in the localization ability between normal hearing and hearing-impaired people be measured

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Dillier, Prof. Dr., Principal Investigator — University of Zurich